CLINICAL TRIAL: NCT02552173
Title: The Relationship Between Operative and Radiologic Stem Version : Which Factors Influence Resultant Stem Version in Primary Total Hip Arthroplasty
Brief Title: The Relationship Between Operative and Radiologic Stem Version
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Hoi Koo, Director, Head of Orthopaedics, Principal Investigator, Professor, Seoul National University Bundang Hospital
Other Study IDs: Ante-002
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Arthroplasty Total Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stem anteversion: intraoperative surgeon's estimation and postopertive CT sacn were taken to measure stem anteversion
  Interventions: Radiation: The Relationship Between Operative and Radiologic Stem Version

INTERVENTIONS:
Radiation: The Relationship Between Operative and Radiologic Stem Version — intraopertive surgeon's estimation and postoperative CT scan

SUMMARY:
Investigators prospectively evaluate the accuracy of intraoperative stem anteversion in 40consecutive total hip arthroplasties.

DETAILED DESCRIPTION:
In all hips, investigators measure femoral stem anteversion postoperatively with three-dimensional computed tomography reconstruction of the femur, using both the distal femoral epicondyles and the posterior femoral condyles to determine the femoral diaphyseal plane. And investigators compare the surgeon's estimate of intraoperative stem version and stem version of CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Investigators recruited 40 consecutive patients who underwent THR between October 2015 and December 2015

Exclusion Criteria:

* patients who could not extend the hip because of a residual flexion contracture.

who had a flexion contracture of the knee or who could not flex the hip to 90° even after THR were excluded because participants could not adopt the posture required for the particular radiographs and CT scans.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Between October 2015 and December 2015, 40 consecutive patients who underwent primary cementless total hip arthroplasty agreed to undergo a postoperative computed tomography scan.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Intraopertive surgeon's estimation and postoperative CT scan were taken to measure stem anteversion | postoperative 4days

SECONDARY OUTCOMES:
The correlation between stem anteversion of intraopertive surgeon's estimation and stem version postoperative CT scan | postoperative 4days
  to determine ICC(intraclass coefficient, correlation coefficient)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, professor, Principal Investigator — Director, Head of Orthopaedics, Seoul National university Bundang Hospital
Locations (1):
- Seoul national University Bundang Hospital, Seongnam-si, Gyeounggi-do, South Korea